CLINICAL TRIAL: NCT03554694
Title: Does Stimulating Friendly Gut Bacteria Improve Brain Function and Behaviour?
Brief Title: Gut-brain Axis, Brain Function, and Behaviour.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Oxford Health Biomedical Research Centre (OH BRC) support scheme (Unknown); Wellcome Centre for Integrative Neuroimaging (Unknown); Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: R52324_RE001
Record Dates: First submitted 2018-05-09; First posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Prebiotics; Anxiety; Humans; Magnetic Resonance Imaging; Decision Making; Emotion; Cortisol
MeSH Terms: conditions — Anxiety Disorders | interventions — Prebiotics; maltodextrin

STUDY DESIGN:
Intervention Model Description: Crossover Assignment Randomised Double-blind Cross-over design with 4-6 weeks of prebiotics intervention and 4-6 weeks of placebo intervention. The first intervention phase will be followed by a 3 week wash-out period prior to the second intervention phase.d.
Who Masked: Participant, Investigator
Masking Description: Both intervention and placebo products are similar in colour, texture, and taste. A third party, independent of the daya-to-day research coordinator, will randomise treatments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Start with prebiotics (Experimental): Half of the participants start with prebiotics, followed by a testing period. After a wash-out period they will continue with placebo followed by a testing period.
  Interventions: Dietary Supplement: Prebiotics
- Start with placebo (Experimental): Half of the participants start with placebo, followed by a testing period. After a wash-out period they will continue with prebiotics followed by a testing period.
  Interventions: Dietary Supplement: Maltodextrin (placebo)

INTERVENTIONS:
Dietary Supplement: Prebiotics — Galactooligosaccharides (GOS) (prebiotics) will be consumed by the participants for 4-6 weeks
  Arms: Start with prebiotics
Dietary Supplement: Maltodextrin (placebo) — Maltodextrin (placebo) will be consumed by the participants for 4-6 weeks
  Arms: Start with placebo

SUMMARY:
The aim is to test if dietary supplementation with prebiotics reduces measures of anxiety in healthy human participants with high self-reported levels of anxiety. Study will test for an effect on behavioural, neuroendocrine and brain imaging markers of anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Trait anxiety levels > 40 on STAI trait inventory
* Participant is willing and able to give informed consent for participation in the study
* Not currently taking any psychoactive medications

Exclusion Criteria:

* Pregnant participants
* No contraindications to prebiotic administration
* Antibiotic, probiotics and/or prebiotic treatment in at least the two previous months.
* Participants who are taking any other food supplements that, in the opinion of the Investigators, may affect the results.
* Participants who are taking any medications that, in the opinion of the Investigators, may affect the results.
* Any significant change in diet which, at the discretion of the Investigators, may affect the results.
* Participants who have recently participated in another research trial which, at the discretion of the Investigators, may affect the results.
* A history of dementia, traumatic brain injury or stroke.
* Anyone who is unable to perform the behavioural tasks.
* Current use of any psychoactive medication.
* Current use of psychological treatment.
* Anyone who does not have adequate understanding of English, sufficient to give informed consent.
* Any person who has a history of drug abuse or a previous history of a neurological, or has a history of neurosurgical procedure is excluded as they may be at increased risk of epilepsy and data collected may be influenced by their condition.
* Anyone with any metal implants or implantable device would be excluded from any brain imaging studies as indicated by the MRI safety screening form.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-05-06 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Cortisol awakening response (CAR) | Cortisol awakening responses will be measured at the end of the first intervention phase (4-6 weeks after study entry) and at the end of the second intervention phase (11-15 weeks post study entry).
  CAR, a marker of stress responsivity, should be decreased after taking prebiotics compared to placebo (as previously found in non-anxious participants in Schmidt et al., 2015, Psychopharmacology)
Brain imaging (BOLD fMRI activity) in amygdala and cortical regions | Brain imaging will be measured at the end of the first intervention phase (4-6 weeks after study entry) and at the end of the second intervention phase (11-15 weeks post study entry).
  Brain imaging (BOLD fMRI activity) in amygdala and cortical regions Will provide neural measures of threat reactivity. We predict decreased amygdala and/or increased parietal-prefrontal brain activity after prebiotics compared to placebo, indicating an anxiolytic-like profile (fearful -neutral face trials in the low load condition) (as in Bishop et al, 2007 and Ironside et al, 2017)

SECONDARY OUTCOMES:
Changes in gut microbiome | Changes in the microbiome will be measure using a single stool/faecal sample at four time points: baseline (0 weeks), following first intervention (4-6 weeks), following washout (7-9 weeks), and following the second intervention (11-15 weeks).
  Availability of specific bacteria in microbiome will change as function of prebiotics and not during placebo. The change will be measured at the start of each intervention compared to the end of each intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jacinta O'Shea, PhD, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The study staff will ensure that the participants' data are safeguarded. The study will comply with the Data Protection Act, which requires personal data to be anonymised as soon as it is practical to do so. Students and collaborators may be given access to fully anonymized data under the supervision of the named investigators. Some peer-reviewed journals require submission of anonymised data that may also be uploaded to other data sharing initiatives. Access may be given to responsible members of the University of Oxford for the purposes of monitoring or audit. The participants' consent will be sought if this is to occur.

REFERENCES:
- [Background] Schmidt K, Cowen PJ, Harmer CJ, Tzortzis G, Errington S, Burnet PW. Prebiotic intake reduces the waking cortisol response and alters emotional bias in healthy volunteers. Psychopharmacology (Berl). 2015 May;232(10):1793-801. doi: 10.1007/s00213-014-3810-0. Epub 2014 Dec 3. PMID 25449699
- [Background] Bishop SJ, Jenkins R, Lawrence AD. Neural processing of fearful faces: effects of anxiety are gated by perceptual capacity limitations. Cereb Cortex. 2007 Jul;17(7):1595-603. doi: 10.1093/cercor/bhl070. Epub 2006 Sep 6. PMID 16956980